CLINICAL TRIAL: NCT04400552
Title: Perioperative Oral Nutrition Supplementation in Malnourished Surgical Cancer Patients- A Randomized Controlled Trial
Brief Title: Perioperative Oral Nutrition Supplementation in Malnourished Surgical Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Collaborators: Kotra Pharma (M) Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Winnie Chee, Principal Investigator, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMU R204/2017
Record Dates: First submitted 2020-04-28; First posted 2020-05-22 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Cancer of Breast; Cancer Colon
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ONS Pre-op + ONS Post-op (Active Comparator): Oral nutrition supplementation (ONS) pre-operatively and post-operatively up to being discharged from hospital
  Interventions: Dietary Supplement: ONS Pre-op + ONS Post-op
- ONS Pre-op + ONS Post-op + ONS Post-op 3 months (Active Comparator): Oral nutrition supplementation (ONS) pre-operatively, post-operatively up to being discharged from hospital and an extended oral nutrition supplementation post-operatively up to 3 months
  Interventions: Dietary Supplement: ONS Pre-op + ONS Post-op + ONS Post-op 3 months
- Usual intake Pre-op + ONS Post-op (Active Comparator): Follow a meal plan of 2000 kcal / day using conventional foods and oral nutrition supplementation (ONS) post-operatively up to being discharged from hospital
  Interventions: Dietary Supplement: Usual intake Pre-op + ONS Post-op

INTERVENTIONS:
Dietary Supplement: ONS Pre-op + ONS Post-op — Participants will consume the oral nutrition supplementation (ONS) in addition to normal diet for 14 days pre-operatively and post-operatively up to participants being discharged from the hospital.
  Arms: ONS Pre-op + ONS Post-op
Dietary Supplement: ONS Pre-op + ONS Post-op + ONS Post-op 3 months — Participants will consume the oral nutrition supplementation (ONS) in addition to normal diet for 14 days pre-operatively, post-operatively up to participants being discharged from the hospital and an extended oral nutrition supplementation post-operatively up to 3 months.
  Arms: ONS Pre-op + ONS Post-op + ONS Post-op 3 months
Dietary Supplement: Usual intake Pre-op + ONS Post-op — Participants will follow a meal plan of 2000 kcal / day using conventional foods for 14 days pre-operatively and consume oral nutrition supplementation (ONS) in addition to normal diet post-operatively up to participants being discharged from the hospital
  Arms: Usual intake Pre-op + ONS Post-op

SUMMARY:
The aim of this study is to evaluate the effectiveness of perioperative oral nutrition supplementation (ONS) on nutritional status in malnourished cancer patients undergoing elective surgery.

The hypothesis is pre-operative ONS feeding in malnourished surgical cancer patients is effective on improving nutritional status. An extended period of 3 months post-operative ONS feeding is effective on improving nutritional status as compared to ONS feeding post-operatively during hospital stay only. Perioperative feeding is effective on improving secondary outcomes such as sleep quality, post-operative complications and length of hospital stay.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effectiveness of perioperative oral nutrition supplementation (ONS) on nutritional status in malnourished cancer patients undergoing elective surgery.

The specific objectives are:

1. To evaluate the baseline nutritional status of cancer patients undergoing elective surgery
2. To evaluate the effectiveness of pre-operative ONS feeding on nutritional status in malnourished surgical cancer patients
3. To evaluate the effectiveness of an extended 3 months post-operative ONS feeding after discharge versus ONS feeding only post-operatively during hospital on nutritional status
4. To evaluate secondary outcomes of perioperative feeding such as sleep quality, post-operative complications and length of hospital stay

Study Design: This is a randomised-controlled-open label-parallel group(s)-trial which will be conducted on malnourished cancer patients undergoing elective surgery.

Study duration: The participation duration for each participant is 4 months. The completion of the study will take around 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from all ethnicity
* 25 to 65 years
* BMI not less than 18.0 kg/m²
* Cancer patients who are confirmed with elective surgery whose co-morbidities are stabilized based on the ASA Physical Status Classification System ASA Class 1 and 2
* Fulfil at least two characteristics of AND/ ASPEN Diagnosis of Malnutrition These characteristics are insufficient energy intake, weight loss, loss of muscle mass, loss of subcutaneous fat, localized or generalized fluid accumulation and diminished functional status as measured by handgrip strength.

Exclusion Criteria:

* Patients who require enteral or parenteral feeding
* Pregnant or lactating
* On chemotherapy or radiotherapy
* Total gastrectomy or ileostomy
* Metastasized cancer, upper gastrointestinal cancer, terminal diseases, decompensated liver or renal disease, major concurrent metabolic problem such as uncontrolled diabetes, dementia
* On regular steroids prescription

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Change from baseline body weight at 4 months
  Anthropometry measurement
Change in body mass index (BMI) | Change from baseline body mass index (BMI) at 4 months
  Anthropometry measurement
Change in serum albumin level | Change from baseline serum albumin level at 4 months
  Serum albumin is an indicator of protein stores to assess nutritional status
Change in serum pre-albumin level | Change from baseline serum pre-albumin level at 4 months
  Serum pre-albumin is an indicator of protein stores to assess nutritional status

SECONDARY OUTCOMES:
Change in handgrip force | Change from baseline handgrip force at 4 months
  Handgrip force is a measure of handgrip strength by dynamometer
Change in muscle mass | Change from baseline muscle mass at 4 months
  Muscle mass reported in kilogram is measured by bioelectrical impedance analyser
Change in fat mass | Change from baseline fat mass at 4 months
  Fat mass reported in kilogram is measured by bioelectrical impedance analyser
Change in serum transferrin level | Change from baseline serum transferrin level at 4 months
  Serum transferrin is a measure of nutritional status
Change in hemoglobin level | Change from baseline hemoglobin level at 4 months
  Serum hemoglobin is a measure of nutritional status
Change in high sensitivity c-reactive protein (HsCRP) level | Change from baseline high sensitivity c-reactive protein (HsCRP) level at 4 months
  High sensitivity c-reactive protein (HsCRP) is a measure of inflammatory status
Change in Interleukin-6 (IL-6) | Change from baseline Interleukin-6 (IL-6) at 4 months
  Interleukin-6 (IL-6) is a measure of inflammatory status
Change in salivary cortisol level | Change from baseline salivary cortisol level at 4 months
  Salivary cortisol level is a biological marker of stress reaction
Change in energy intake | Change from baseline energy intake at 4 months
  Energy intake reported in calories is a dietary measure to assess nutritional status
Change in protein intake | Change from baseline protein intake at 4 months
  Protein intake reported in gram is a dietary measure to assess nutritional status
Change in Pittsburgh Sleep Quality Index (PSQI) scores | Change from baseline Pittsburgh Sleep Quality Index (PSQI) scores at 4 months
  Pittsburgh Sleep Quality Index (PSQI) scores range from 0-42.Higher scores indicate poorer sleep quality
Presence of post-surgical complications | Change from baseline post-surgical complications at 3 months
  Post-surgical complications are indicated by presence of wound infection, chest infection and use of antibiotics, responses are either yes or no
Length of hospital stay | Up to 5 days
  Number of days participants are admitted into the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Winnie SS Chee, PhD, Principal Investigator — IMU University, Malaysia
Locations (1):
- International Medical University, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong TX, Chen ST, Ong SH, Shyam S, Kandasami P, Chee WSS. Study protocol for an open labelled randomised controlled trial of perioperative oral nutrition supplement in breast and colorectal cancer patients undergoing elective surgery. Trials. 2021 Nov 3;22(1):767. doi: 10.1186/s13063-021-05716-5. PMID 34732233